CLINICAL TRIAL: NCT00850213
Title: Registro Redes - Evaluación Del Comportamiento clínico y Del Coste Del Stent Coronario Endeavor Resolute de Medtronic "en el Mundo Real" en España
Brief Title: Assessment of Clinical Performance and Costs of the Endeavor Resolute Stent "in Real Life" in Spain.
Acronym: REDES
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: MDT-REDES1.7
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2012-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Endeavor Resolute Stent: Patients implanted with the Medtronic Endeavor Resolute stent
  Interventions: Device: Endeavor Resolute Stent

INTERVENTIONS:
Device: Endeavor Resolute Stent — Single implantation
  Other Names: Medtronic Endeavor Resolute Coronary Stent System

SUMMARY:
The Redes registry is set up to document the overall clinical performance and costs of the Endeavor Resolute coronary stent in a "real life" subject population of 450 patients that require a stent in Spain. Primary objectives are the overall cost for patients during initial hospitalization and at 1-year follow-up, as well as the MACE rate at 30 days, 6 months and 12 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >18 years old
* Subject has agreed to participate in the study by signing the "Patient Informed Consent" and/or has authorized the collection and disclosure of their personal health information by signing the "Patient Data Collection Form".
* There is an indication for a drug-eluting stent and a clinical decision to use Endeavor Resolute in all the lesions found.
* Subject is able and willing to co-operate and to comply with the study protocol and undergo follow-up requirements.

Exclusion Criteria:

* Subject is a childbearing or breastfeeding female.
* Subject has a known hypersensitivity or allergy to acetylsalicylic acid, heparin, clopidogrel, ticlopidine, drugs such as zotarolimus, rapamycin, tacrolimus, sirolimus or other similar drugs, or any other analog or derivative drug, cobalt, chrome, nickel, molybdenum or contrast media.
* Subject has a contraindication to anticoagulants and/or antiplatelets.
* Subject's lesion might prevent proper balloon inflation during angioplasty.
* Primary or rescue angioplasty.
* Subject has one or more drug-eluting stents other than Endeavor Resolute in other lesions.
* Intention for elective treatment with other drug-eluting stent other than Endeavor Resolute.
* Current medical condition is associated with a life expectancy ≤ 12 months.
* Subject is participating in another investigational drug or device study and has not completed the follow-up required for that study at least 30 days prior to signing the consent form in this study. Subject can only be enrolled once in this study.
* Subject has a medical condition preventing follow-up as established in the protocol or limiting participation in this study.
* Subject cannot guarantee follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for an Endeavor Resolute coronary stent. The study will include all consecutive patients who are appropriate candidates for at least one Endeavor Resolute stent in at least one target lesion after angiography.
Sampling Method: Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Overall patient cost | During initial hospitalization and at 12 month follow-up
Number of major adverse cardiac events (MACE) | 30 days, 6 months and 1 year

SECONDARY OUTCOMES:
Rate of stent thrombosis (according to ARC criteria, defined as definite/confirmed, probable and possible) | 12 Months
Target Lesion Revascularization (TLR) | 12 Months
Procedure, device and lesion success rate | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: José Moreu Burgos, Dr., Principal Investigator — Hospital Virgen de la Salud
Locations (6):
- Spain (6):
  - Hospital Juan Canalejo, A Coruña
  - Hospital General de Alicante, Alicante
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital de León, León
  - Hospital Cínico Universitario de Málaga, Málaga
  - Hospital Virgen de la Salud, Toledo